CLINICAL TRIAL: NCT03507322
Title: Ultrasound Study Through Uterine Texturization to Predict Pregnancy After Blastocyst Transfer in Patients Undergoing Hormone Replacement Therapy (HRT) Cycles With Donor Oocytes
Brief Title: Ultrasound Study by Texturization as a Predictor of Pregnancy in Oocyte Donation Programs
Acronym: TEXTUGEST
Status: Withdrawn | Type: Observational
Why Stopped: Clinic management decided to cancel the study for priority reasons
Sponsor: Vida Recoletas Sevilla (Other)
Responsible Party: Sponsor
Other Study IDs: 1605-SEV-034-IR
Record Dates: First submitted 2017-11-10; First posted 2018-04-25 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Infertility
Keywords: texturization; pregnancy rate; oocyte donation; 2D ultrasound; 3D ultrasound; assisted reproductive technology (ART)
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ultrasound texturization: Application of ultrasound texturization (2D/3D ultrasound scanning)
  Interventions: Other: Ultrasound texturization

INTERVENTIONS:
Other: Ultrasound texturization — Along several visits to the clinic, the patients will be subjected to 2D/3D ultrasound scanning.

SUMMARY:
This study is focused on analysing the application of ultrasound scanning techniques as new biomarkers in reproductive medicine. Those biomarkers are based on the analysis of ultrasound texture in different areas of uterine tissue, using 2D/3D ultrasound scanning. Investigators will use the algorithm Text® to analyse the ultrasound texture of the endometrium and myometrium. The aim of the project is to study if it is possible to obtain measurable, objective and reproducible data in healthy volunteers which can be used to predict pregnancy and determine the best moment to perform embryo transfer in assisted reproductive technology (ART) cycles

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18 and 30 kg/m2
* Not taking the contraceptive pill in a previous cycle
* Non-pregnant: beta human chorionic gonadotropin (HCG) test with negative result at the beginning of the study)
* No previous history of inflammatory diseases, circulatory diseases, abdomen or pelvic diseases
* Physical gynecological exploration without pathological findings
* Gynecological ultrasound study of the uterus with a normal result

Exclusion Criteria:

* Ultrasound studies with technical defects in image acquisition
* Simultaneous participation in other studies
* Previous participation in other study which can affect the results of the present study

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Infertile women undergoing IVF/ICSI treatment
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2018-09-10 (Actual); Study Completion 2018-09-10 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | Around 5-6 weeks after embryo transfer
  Detection of gestational sac through ultrasound scanning indicating clinical pregnancy
Biochemical miscarriage rate | Up to one month after embryo transfer
  Interruption of pregnancy after a positive result in the beta HCG test
Clinical miscarriage rate | Up to 20 weeks after embryo transfer
  Interruption of pregnancy after confirming clinical pregnancy using ultrasound scanning
Chemical pregnancy rate | Around 14 days after embryo transfer
  Positive result in beta HCG test indicating pregnancy
beta HCG level | Around 14 days after embryo transfer
  Level of beta HCG in the test performed to detect pregnancy

CONTACTS AND LOCATIONS:
Locations (1):
- IVI Sevilla, Seville, Spain